CLINICAL TRIAL: NCT05052190
Title: Improving Influenza Vaccination Delivery Across a Health System by the Electronic Health Records Patient Portal RCT 4
Brief Title: Patient Portal Flu Vaccine Reminders_RCT 4
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IT error which contaminated study arms
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Executive Vice Chair, Clinical Research, UCLA David Geffen School of Medicine, Dept of Pediatrics, University of California, Los Angeles, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-001889-AM-00015; R01AI135029-04 (NIH)
Record Dates: First submitted 2021-08-31; First posted 2021-09-22 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Influenza; Respiratory Tract Infections
Keywords: Reminder Recall (R/R); Influenza Vaccine; Electronic Health Record; Text Message; Vaccine
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Pragmatic comparative effectiveness trial with a standard-of-care control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Text Message R/R with Direct Appointment Schedule Link (Active Comparator): Participants in this arm will receive up to 3 R/R messages by text. R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Interventions: Behavioral: Text Message R/R with Direct Appointment Schedule Link
- Text Message R/R without Direct Appointment Schedule Link (Active Comparator): Participants in this arm will receive up to 3 R/R messages by text with no link to schedule an appointment.
  Interventions: Behavioral: Text Message R/R without Direct Appointment Schedule Link
- Text Message R/R with Direct Appointment Schedule Link + text Pre-Appointment Reminder (Active Comparator): Participants in this arm will receive up to 3 R/R messages by text. R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment. Participants will receive a Pre-Appointment Reminder via text when they schedule a visit during the study period.
  Interventions: Behavioral: Text Message R/R with Direct Appointment Schedule Link; Behavioral: Text Pre-Appointment Reminder
- Text Message R/R without Direct Appointment Schedule Link + Text Pre-Appointment Reminder (Active Comparator): Participants in this arm will receive up to 3 R/R messages by text. R/R message will be sent without a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment. Participants will receive a Pre-Appointment Reminder via text when they schedule a visit during the study period.
  Interventions: Behavioral: Text Message R/R without Direct Appointment Schedule Link; Behavioral: Text Pre-Appointment Reminder
- Portal Message R/R with Direct Appointment Schedule Link (Active Comparator): Participants in this arm will receive up to 3 R/R messages by portal. R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Interventions: Behavioral: Portal Message R/R with Direct Appointment Schedule Link
- Portal Message R/R without Direct Appointment Schedule Link (Active Comparator): Participants in this arm will receive up to 3 R/R messages by portal. R/R message will be sent without a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Interventions: Behavioral: Portal Message R/R without Direct Appointment Schedule Link
- Portal Message R/R with Direct Appointment Schedule Link + Portal Pre-Appointment Reminder (Active Comparator): Participants in this arm will receive up to 3 R/R messages by portal. R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment. Participants will receive a Pre-Appointment Reminder advising them to ask their doctor for the flu vaccine at their upcoming appointment via portal when they schedule a visit during the study period.
  Interventions: Behavioral: Portal Message R/R with Direct Appointment Schedule Link; Behavioral: Portal Pre-Appointment Reminder
- Portal Message R/R without Direct Appointment Schedule Link + Portal Pre-Appointment Reminder (Active Comparator): Participants in this arm will receive up to 3 R/R messages by portal. R/R message will be sent without a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment. Participants will receive a Pre-Appointment Reminder advising them to ask their doctor for the flu vaccine at their upcoming appointment via portal when they schedule a visit during the study period.
  Interventions: Behavioral: Portal Message R/R without Direct Appointment Schedule Link; Behavioral: Portal Pre-Appointment Reminder
- No R/R Message or Pre-Appointment Reminder (No Intervention): Participants do not receive any flu vaccine R/R message or Pre-Appointment Reminder advising them to ask their doctor for the flu vaccine at their upcoming appointment during the specified flu season.

INTERVENTIONS:
Behavioral: Text Message R/R with Direct Appointment Schedule Link — Participants in this arm will receive up to 3 R/R messages by text reminding them to get a flu vaccine with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Arms: Text Message R/R with Direct Appointment Schedule Link; Text Message R/R with Direct Appointment Schedule Link + text Pre-Appointment Reminder
Behavioral: Text Message R/R without Direct Appointment Schedule Link — Participants in this arm will receive up to 3 R/R messages by text reminding them to get a flu vaccine without a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Arms: Text Message R/R without Direct Appointment Schedule Link; Text Message R/R without Direct Appointment Schedule Link + Text Pre-Appointment Reminder
Behavioral: Text Pre-Appointment Reminder — Participants will receive a Pre-Appointment Reminder via text when they schedule a visit during the study period advising them to get the flu vaccine at their upcoming appointment.
  Arms: Text Message R/R with Direct Appointment Schedule Link + text Pre-Appointment Reminder; Text Message R/R without Direct Appointment Schedule Link + Text Pre-Appointment Reminder
Behavioral: Portal Message R/R with Direct Appointment Schedule Link — Participants in this arm will receive up to 3 R/R messages by portal. R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Arms: Portal Message R/R with Direct Appointment Schedule Link; Portal Message R/R with Direct Appointment Schedule Link + Portal Pre-Appointment Reminder
Behavioral: Portal Message R/R without Direct Appointment Schedule Link — Participants in this arm will receive up to 3 R/R messages by portal. R/R message will be sent without a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Arms: Portal Message R/R without Direct Appointment Schedule Link; Portal Message R/R without Direct Appointment Schedule Link + Portal Pre-Appointment Reminder
Behavioral: Portal Pre-Appointment Reminder — Participants will receive a Pre-Appointment Reminder via the portal advising them to ask their doctor for the flu vaccine at their upcoming appointment via text when they schedule a visit during the study period.
  Arms: Portal Message R/R with Direct Appointment Schedule Link + Portal Pre-Appointment Reminder; Portal Message R/R without Direct Appointment Schedule Link + Portal Pre-Appointment Reminder

SUMMARY:
This trial is taking place in Los Angeles, CA at clinics within the UCLA Health System.

The study design is a 2x2 nested factorial design. Patients will be randomized into 1) receiving text based reminder messages, 2) portal-based reminder messages or 3) the control group. Patients randomized to the intervention arms will receive reminders if they are due for influenza vaccine.

Nested within the reminder arms (text or portal), we will have 2 additional components for which patients will be randomized separately:

* A direct scheduling link within the reminder letter enabling the patient to schedule an influenza vaccine only visit (direct scheduling link vs. no direct scheduling link).
* A pre-appointment reminder, encouraging patients to ask for their influenza vaccine at their upcoming appointment (pre-appointment reminder encouraging influenza vaccination vs. standard pre-appointment reminder not mentioning influenza vaccination)

Despite the Advisory Committee on Immunization Practices (ACIP) recommendation in 2010 that all people above 6 months of age should receive an annual flu vaccine, vaccination rates remain low: at 6m-4.9 yrs. (70%), 5-17.9 yrs. (56%), 18-64.9 yrs. (38%), and >65 yrs. (63%). The investigators will assess the effectiveness of MyChart R/R messages and text R/R messages as compared to the standard of care control (no messages).

DETAILED DESCRIPTION:
Sub-optimal vaccination rates are a significant problem in the U.S., despite their effectiveness in preventing morbidity and mortality from vaccine-preventable illness. For influenza specifically, annual epidemics of influenza cause substantial morbidity in the U.S. with up to 40,00-80,000 deaths/year and many hospitalizations, emergency and outpatient visits, and significant costs.

Reminder/recall (R/R), sent by phone, mail or other modality, can improve child and adult influenza vaccination rates. However, the majority of pediatric or adult primary care practices do not conduct R/R. Barriers are lack of finances, personnel, and algorithms to identify eligible patients.

A technological breakthrough that might overcome these barriers involves patient portals-- secure, web-based communication systems, embedded within electronic health records (EHRs), for patients and providers to communicate with each other via email and the internet. Portals are used by about half of Americans and half of UCLA patients. Another is text messaging at the health system level.

This randomized controlled trial will assess the effectiveness of reminders messages sent to portal users, encouraging influenza vaccination, on increasing influenza vaccination rates within a health system. Patients will be randomized into three groups: 1) one-third of patients will receive reminder letters via the portal, 2) one-third will receive reminders via text messages sent by the health system and 3) one-third will not receive reminders.

Patients in the reminder arms will be further randomized (separately) for two additional components: 1) direct appointment scheduling and 2) pre-appointment reminders.

Direct scheduling: The convenience of scheduling an appointment for influenza vaccination may increase the likelihood that patients receive an influenza vaccination. Patients receiving reminders will be randomized to receive one of two types of reminder letters: 1) one half will receive flu vaccine reminder letters with a link to the MyChart direct appointment scheduling page and 2) one half will receive flu vaccine reminder message without the direct appointment scheduling link.

Pre-appointment flu reminders: Finally, a missed opportunities for vaccination occurs when patients are eligible for vaccination but are not offered a vaccine at their medical appointment. Pre-appointment reminders, sent in advance of an upcoming appointment, encouraging the patient talk to their doctor about influenza vaccination, may increase the likelihood of that patient receiving a vaccine. Patients will be randomized to one of two groups: 1) one half will receive modified pre-appointment reminders that mention influenza vaccination and 2) one half will receive the standard pre-appointment reminders for an upcoming appointment (no mention of influenza vaccination).

Interventions that apply Behavioral Economics principles in vaccine promotion messaging can increase vaccine receipt. We will include ownership language in the pre-appointment messages. Additionally, the convenience of reminders sent via text and with a Direct Appointment Schedule link included enables patients to self-schedule a flu vaccine only visit, reducing friction for vaccine receipt.

For the primary analysis, the primary outcome will be the patient's end of flu season vaccination status. Intervention effects will be assessed using mixed effects log-binomial models. Models will contain terms for messaging modality (text v. portal v. none), pre-appointment reminders (sent v. not sent), and direct scheduling link (included v. not included).

The R/R text and portal messages (with and without direct scheduling links) and pre-appointment reminders and will all begin in October of 2021.

ELIGIBILITY:
Inclusion Criteria:

* Active Portal Users A patient within the UCLA Health System identified as a primary care patient per an internal algorithm

Exclusion Criteria:

* A patient within the UCLA Health System not identified as a primary care patient per an internal algorithm

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 239567 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MPH, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California LA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text Message R/R With Direct Appointment Schedule Link | Text Message R/R Without Direct Appointment Schedule Link | Text Message R/R With Direct Appointment Schedule Link + Text Pre-Appointment Reminder | Text Message R/R Without Direct Appointment Schedule Link + Text Pre-Appointment Reminder | Portal Message R/R With Direct Appointment Schedule Link | Portal Message R/R Without Direct Appointment Schedule Link | Portal Message R/R With Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | Portal Message R/R Without Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | No R/R Message or Pre-Appointment Reminder
Started | 19975 | 19938 | 19991 | 19950 | 20047 | 20008 | 20061 | 20027 | 79570
Completed | 19975 | 19938 | 19991 | 19950 | 20047 | 20008 | 20061 | 20027 | 79570
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text Message R/R With Direct Appointment Schedule Link | Text Message R/R Without Direct Appointment Schedule Link | Text Message R/R With Direct Appointment Schedule Link + Text Pre-Appointment Reminder | Text Message R/R Without Direct Appointment Schedule Link + Text Pre-Appointment Reminder | Portal Message R/R With Direct Appointment Schedule Link | Portal Message R/R Without Direct Appointment Schedule Link | Portal Message R/R With Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | Portal Message R/R Without Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | No R/R Message or Pre-Appointment Reminder | Total
Number analyzed (Participants) | 19975 | 19938 | 19991 | 19950 | 20047 | 20008 | 20061 | 20027 | 79570 | 239567
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1748 | 1743 | 1737 | 1738 | 1773 | 1794 | 1804 | 1767 | 7083 | 21187
  Between 18 and 65 years | 14222 | 14227 | 14296 | 14093 | 14299 | 14180 | 14263 | 14210 | 56468 | 170258
  >=65 years | 4005 | 3968 | 3958 | 4119 | 3975 | 4034 | 3994 | 4050 | 16019 | 48122
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 11344 | 11251 | 11315 | 11352 | 11426 | 11301 | 11409 | 11405 | 45246 | 136049
  Male | 8627 | 8683 | 8670 | 8597 | 8618 | 8707 | 8647 | 8620 | 34315 | 103484
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown | 4 | 2 | 2 | 1 | 2 | 0 | 2 | 0 | 5 | 18
  Missing | 0 | 2 | 4 | 0 | 1 | 0 | 3 | 2 | 4 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 2179 | 2235 | 2247 | 2207 | 2269 | 2297 | 2325 | 2205 | 8866 | 26830
  Ethnicity: Not Hispanic or Latino | 14630 | 14575 | 14563 | 14628 | 14529 | 14538 | 14523 | 14638 | 58141 | 174765
  Ethnicity: Unknown | 3166 | 3128 | 3181 | 3115 | 3249 | 3173 | 3213 | 3184 | 12563 | 37972
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 55 | 51 | 60 | 60 | 55 | 50 | 42 | 53 | 217 | 643
  Race: Asian | 1888 | 1944 | 1940 | 1850 | 1920 | 1883 | 1944 | 1897 | 7733 | 22999
  Race: Black | 965 | 941 | 950 | 971 | 984 | 976 | 1003 | 946 | 3840 | 11576
  Race: Native Hawaiian or Other Pacific Islander | 38 | 39 | 42 | 32 | 40 | 32 | 39 | 42 | 173 | 477
  Race: White or Caucasian | 10750 | 10779 | 10754 | 10793 | 10580 | 10805 | 10718 | 10729 | 42682 | 128590
  Race: Other | 2717 | 2661 | 2693 | 2683 | 2771 | 2697 | 2693 | 2705 | 10797 | 32417
  Race: Multiracial | 565 | 532 | 552 | 603 | 620 | 572 | 544 | 637 | 2246 | 6871
  Race: Unknown | 2988 | 2975 | 2986 | 2946 | 3060 | 2974 | 3064 | 3008 | 11817 | 35818
  Race: Missing | 9 | 16 | 14 | 12 | 17 | 19 | 14 | 10 | 65 | 176

OUTCOME MEASURES:

1. Primary Outcome: Receipt of the Annual Influenza Vaccine Among Adult and Pediatric Index Patients
Description: Percent of patients with annual influenza vaccination (between 10/1/21 - 4/1/22) among adult and pediatric index patients. Outcomes will be assessed via vaccine data extraction from the electronic health record and external claims and pharmacy data.
  The index patients must also be an active UCLA Health MyChart user (>= 1 login over the last 12 months from 8/1/21, excluding activity on the user's initial profile activation date). Individuals not affiliated with any primary care practice will be excluded from the primary analysis.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Text Message R/R With Direct Appointment Schedule Link | Text Message R/R Without Direct Appointment Schedule Link | Text Message R/R With Direct Appointment Schedule Link + Text Pre-Appointment Reminder | Text Message R/R Without Direct Appointment Schedule Link + Text Pre-Appointment Reminder | Portal Message R/R With Direct Appointment Schedule Link | Portal Message R/R Without Direct Appointment Schedule Link | Portal Message R/R With Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | Portal Message R/R Without Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | No R/R Message or Pre-Appointment Reminder
Number analyzed (Participants) | 19975 | 19938 | 19991 | 19950 | 20047 | 20008 | 20061 | 20027 | 79570
Participants | 8360 | 8495 | 8564 | 8377 | 8055 | 7928 | 8035 | 8075 | 32537

2. Other Pre Specified Outcome: Receipt of the Annual Influenza Vaccine Among Pediatric Index Patients
Description: Percent of patients with annual influenza vaccination (between 10/1/21 - 4/1/22) among pediatric index patients. Outcomes will be assessed via vaccine data extraction from the electronic health record and external claims and pharmacy data.
  The index patients must also be an active UCLA Health MyChart user (>= 1 login over the last 12 months from 8/1/21, excluding activity on the user's initial profile activation date). Individuals not affiliated with any primary care practice will be excluded from the primary analysis.
Time Frame: 6 months - Unable to analyze data due to contaminated study arms
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: We did not collect information regarding adverse events.
Description: We did not collect adverse event information. We monitored whether reminder recall through the portal and text was effective at increased influenza vaccination rates. Because influenza vaccination is recommended by the Advisory Committee on Immunization Practices and is part of the U.S. recommended vaccine schedule, we did not collect adverse event data.
Arm/Group | Text Message R/R With Direct Appointment Schedule Link | Text Message R/R Without Direct Appointment Schedule Link | Text Message R/R With Direct Appointment Schedule Link + Text Pre-Appointment Reminder | Text Message R/R Without Direct Appointment Schedule Link + Text Pre-Appointment Reminder | Portal Message R/R With Direct Appointment Schedule Link | Portal Message R/R Without Direct Appointment Schedule Link | Portal Message R/R With Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | Portal Message R/R Without Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | No R/R Message or Pre-Appointment Reminder
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Errors occurred with the text messaging component of our studying meaning that over half of the cohort that was randomized to receive the intervention did not receive the allocated messages. For this reason, our study team terminated the study early and had no intention of ever publishing these results but instead planned to repeat the trial correctly. Outcome results reported are not valid and have not been published

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT05052190/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT05052190/SAP_001.pdf